CLINICAL TRIAL: NCT01779895
Title: Effect of Probiotic Lactobacillus Paracasei NCC2461 on House Dust Mite Allergy
Brief Title: Probiotic Administration and Perennial Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12.18.MET
Record Dates: First submitted 2013-01-22; First posted 2013-01-30 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Dust mite; Perennial allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NCC2461 (Active Comparator): probiotic blended in maltodextrin powder to be taken daily
  Interventions: Dietary Supplement: Lactobacillus paracasei probiotic strain
- Placebo (Placebo Comparator): maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei probiotic strain
  Arms: NCC2461
Dietary Supplement: Placebo — maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of a probiotic strain in improving the quality of life in adult subjects suffering from perennial allergic rhinit.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 20-65 years old
* Confirmed allergy (allergic rhinitis) to dust mite for more than 2 years, as determined by anamnesis and by a miniRQLQ of ≥ 1
* Positive Skin prick testing measure greater than 3mm wheal diameter to the dermatophagoides pteronyssinus species of house dust mite extract
* Body Mass Index 19-29
* Having obtained his/her informed consent

Exclusion Criteria:

* Anemia
* Allergy to any food or medication
* Asthma
* Family history of congenital immunodeficiency or chronic consumption (more than one week at Screening) of immunosuppressive or anti-inflammatory treatments
* Ongoing treatment with antibiotics or undergoing allergen immunotherapy at Screening
* Consumption of probiotic and other dietary nutritional interventions
* More than 2 drinks/day alcohol consumption or use of illicit drugs
* Pregnant women
* Subjects with expected low compliance
* Blood donation in the past month or planning to donate blood until a month after the end of the study
* Currently participating or having participated in another interventional clinical trial during the last four weeks prior to the beginning the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Quality of life, measured by a validated mini rhinoconjunctivitis quality of life questionnaire (MiniRQLQ) | 8 weeks
  Compared over 8 weeks between the two treatment groups

SECONDARY OUTCOMES:
Level of pro-inflammatory cytokines in ex-vivo stimulated whole blood cells | Measured 3 times: at the start of product intake, after 4 weeks and after 8 weeks
Basophil activation in ex-vivo stimulated whole blood cells | Measured 3 times: at the start of product intake, after 4 weeks and after 8 weeks
Total Nasal Symptom Score (TNSS), Total Ocular Symptom Score (TOSS), Medication score | Measured weekly for the 8 weeks of product intake
Level of Specific Immunoglobulin E | Measured 2 times: at the start of product intake and after 8 weeks
Frequency of adverse events | during the 8 weeks of product intake

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, Principal Investigator — Nestlé Research Centre
Locations (1):
- Metabolic Unit, Nestlé Research Centre, Lausanne, Switzerland